CLINICAL TRIAL: NCT05162300
Title: An Open Label Cosmetic Study to Evaluate the Safety and Efficacy of the Same-day Treatment of VI Peel® and Botox® for the Correction of Sun Damage, Fine Lines, and Wrinkles on the Face
Brief Title: Same-Day Combination of VI Peel and Botox for Correction of Sun Damage, Fine Lines and Wrinkles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vitality Institute Medical Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-VITA-101
Record Dates: First submitted 2021-11-18; First posted 2021-12-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Photoaging; Wrinkle; Sun Damaged Skin
Keywords: Botox; VI Peel; Wrinkles; Sun Damage
MeSH Terms: interventions — Botulinum Toxins; Pharmaceutical Preparations; Botulinum Toxins, Type A; Tooth Exfoliation; Neurotoxins; Chemexfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Group A (Experimental): Subjects will be given the same-day combination of VI Peel (Procedure) and Botox Cosmetic (Botulinum Toxin) (Drug). Botox will be administered via intramuscular injection via package insert to Glabella, Forehead and Crows Feet. Dosage will follow package insert guidelines.
  The two interventions will be administered once at the start of the study, subsequent study visits will focus on assessment and evaluation.
  Interventions: Combination Product: Same Day Intervention of VI Peel (Procedure) and Botulinum Toxin (Drug)

INTERVENTIONS:
Combination Product: Same Day Intervention of VI Peel (Procedure) and Botulinum Toxin (Drug) — Same-Day combination of VI Peel applied to the full face, followed by Botox injection per label to the face.
  Other Names: Botox; VI Peel; Neurotoxin; Chemical Peel

SUMMARY:
This study is being conducted to improve standards of care in the cosmetic treatment of sun damage, fine lines, and wrinkles. VI Peels® and Botox® have been used cosmetically to improve patient concerns as monotherapies. This study seeks to confirm that the same-day combination creates no additional side-effects and furthermore that patient satisfaction is heightened as a result.

DETAILED DESCRIPTION:
This study seeks to utilize the mechanisms of action of both products to simultaneously address fine lines and wrinkles. VI Peels contain a synergistic blend of acids that produce keratolytic and kerato-coagulation qualities focused on desquamation and cellular renewal. The VI Peel blend contains Trichloroacetic Acid, Phenol, Salicylic Acid, Retinoic Acid and Ascorbic Acid. Botox containing Botulinum toxin type A is a purified substance, derived from a bacterium that block muscular nerve signals temporarily preventing the muscular contraction and subsequent wrinkle formation.

The expected benefit of this investigational combination include improvements to Standards of Care in relation to treatment of the cosmetic patient by establishing safety of the combination treatment, improving patient outcomes by simultaneously addressing sun damage, fine lines, and wrinkles through dual mechanisms, and overall improvement to patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Female and Males subjects of any race
2. Ages 30-70 Years old
3. Subjects who can read, understand, and sign the Informed Consent Form.
4. Subjects willing and able to comply with all study requirements, including return visits and photographs (eyes censored or uncensored).

Exclusion Criteria:

1. Is pregnant or lactating
2. Has an active infection on their face (excluding acne)
3. Has used Isotretinoin (Accutane) within the last six months
4. Has had chemotherapy or radiation treatments within the last six months
5. Has a history of neuromuscular disorders
6. Has a history of bleeding disorders
7. Has an allergy to albumin
8. Has an allergy to Aspirin
9. Has an allergy to Phenol
10. Has received the following treatments in the last 6 months:

    botulinum toxin, soft tissue filler, medium to deep chemical peel, ablative laser, radio frequency treatment, ultrasound device treatment, non-ablative laser treatment
11. Is planning on receiving in the next 1months: soft tissue filler, medium to deep chemical peel, ablative laser, radio frequency treatment, ultrasound device treatment, nonablative laser treatment
12. Is unable to understand the protocol or to give informed consent
13. Not willing to comply with all study requirements including return visits and photographs (eyes censored or uncensored)
14. Has been diagnosed or is displaying COVID-19 symptoms -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 7 (+/- 3)
  To establish safety of the same-day combination of VI Peel & Botox, the study will measure the rate and occurrence of Adverse Events as compared to a stand-alone treatment of Botox.
  Rate and occurrence of Botox as a stand-alone intervention will be based off of the package insert indicating each Adverse Event

SECONDARY OUTCOMES:
Change to Facial Wrinkle Severity | Baseline, 7 (+/- 3) Days after Intervention, and 30 Days after Intervention
  Overall improvements to fine lines and wrinkles will be measured using the Facial Wrinkle Severity Scale described below.
  Facial Wrinkle Severity Scale (FWSS) Grade 0 = no wrinkles; Grade 1 = mild wrinkles; Grade 2 = moderate wrinkles; and Grade 3 = severe wrinkles.
  Principal investigator will rate and measure subject on enrollment into the study, will grade again at Day 7 (+ / - 3) and again at Day 30.
Change to Uniformity of Pigment | Baseline, 7 (+/- 3) Days after Intervention, and 30 Days after Intervention
  Overall improvements to pigment will be measured using the Uniformity of Pigment Scale described below.
  Uniformity of Pigment; Grade 0 = Uniform, Grade 1 = mild, Grade 2 = moderate, Grade 3 = moderate to severe, Grade 4 = Severely Ununiform.
  Principal investigator will rate and measure subject on enrollment into the study, will grade again at Day 7 (+ / - 3) and again at Day 30.
Change to | Baseline, 7 (+/- 3) Days after Intervention, and 30 Days after Intervention
  Overall improvements to Skin Tone will be measured via the Skin Tone grading scale below.
  Skin Tone; Grade 0 = Clear and Radiant, Grade 1 = Mild Irregularities, Grade 2 = Moderate Irregularities, Grade 3 = Moderate to Severe Irregularities, Grade 4 = Severe Irregularities, ie. Sallow, Dull.
  Principal investigator will rate and measure subject on enrollment into the study, will grade again at Day 7 (+ / - 3) and again at Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Roberts, MD, Principal Investigator — Principal Investigator
Locations (1):
- Dr. Wendy E. Roberts, MD, Rancho Mirage, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: MedlinePlus: Botox Cosmetic Overview — https://medlineplus.gov/botox.html
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks